CLINICAL TRIAL: NCT05472155
Title: SUCTIONING AT BIRTH WITH BULB SYRINGE OR SUCTION CATHETER: A RANDOMIZED CONTROLLED TRIAL
Acronym: NEOSUC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Padova (Other)
Collaborators: Doctors with Africa - CUAMM (Other)
Responsible Party: Principal Investigator, Daniele Trevisanuto, Associate Professor, University Hospital Padova
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NEOUNIPD3(2022)
Record Dates: First submitted 2022-07-21; First posted 2022-07-25 (Actual); Last update posted 2023-12-05 (Actual); Status verified 2023-12

CONDITIONS: Neonatal Resuscitation

STUDY DESIGN:
Masking Description: Masking is not possible due to the study design. Only statistician who will perform the analysis will be blind to the arm allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Oropharyngeal suctioning with a bulb syringe (Experimental): Newborn infants who have obvious obstruction to spontaneous breathing or who require positive pressure ventilation immediately after birth will be suctioned with a bulb syringe
  Interventions: Device: Bulb syringe
- Oropharyngeal suctioning with a suction catheter (Active Comparator): Newborn infants who have obvious obstruction to spontaneous breathing or who require positive pressure ventilation immediately after birth will be suctioned with a suction catheter
  Interventions: Device: Suction catheter

INTERVENTIONS:
Device: Bulb syringe — Suctioning with a bulb syringe
  Arms: Oropharyngeal suctioning with a bulb syringe
Device: Suction catheter — Suctioned with a suction catheter
  Arms: Oropharyngeal suctioning with a suction catheter

SUMMARY:
This study is designed to compare two different methods of oropharyngeal suctioning (with bulb syringe or suction catheter) in newborn infants at birth.

DETAILED DESCRIPTION:
Objective of the study: This trial aims to compare two different methods of oropharyngeal suctioning (with bulb syringe or suction catheter) in newborn infants needing suctioning at birth.

Primary outcome measure: Oxygen saturation during the first 10 minutes of life.

Study design: This is a single center, prospective, randomized clinical trial comparing two different methods of oropharyngeal suctioning (with bulb syringe or suction catheter) in newborn infants needing suctioning at birth.

Setting: The study is conducted at the St. Luke Catholic Hospital in Wolisso (Ethiopia), which is a level III hospital with around 3,600 deliveries per year.

Immediately after birth, all infants needing suctioning are randomized to receive suctioning with bulb syringe or suction catheter. All resuscitative procedures are performed following the Helping Babies Breathe algorithm. An external observer, not involved in the care of the newborn, is responsible of the positioning the probe of the pulse oximeter and the collection of the data.

We aim to enroll 60 neonates.

ELIGIBILITY:
Inclusion Criteria:

* inborn infants (and)
* need for suctioning at birth (and)
* parental consent

Exclusion Criteria:

* Major congenital malformations
* Parental refusal to participate in the study

Ages: 1 Minute to 2 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2022-07-21 (Actual); Primary Completion 2022-10-30 (Actual); Study Completion 2022-10-30 (Actual)

PRIMARY OUTCOMES:
Oxygen saturation during the first 10 minutes of life | 10 minutes
  Preductal oxygen saturation will be measured by a pulse-oxymeter during the first 10 minutes of life

SECONDARY OUTCOMES:
Heart rate during the first 10 minutes of life | 10 minutes
  Heart rate will be monitored by a pulse-oxymeter during the first 10 minutes of life
Neonates with heart rate >100 beats per minute at 5 minutes | 5 minutes
  Number (percentage) of neonates with heart rate >100 bpm at 5 minutes
Episodes of bradycardia in the first 10 minutes of life | 10 minutes
  Episodes of bradycardia will be defined as heart rate <100 beats per minute in the first 10 minutes of life
Neonates with saturation >80% at 5 minutes | 5 minutes
  Number (percentage) of neonates with saturation >80% at 5 minutes
Time for achieving transcutaneous saturations >90% | 30 minutes
  Time needed for achieving transcutaneous saturations >90 from birth
Face-mask ventilation | 10 minutes
  Number (percentage) of infants who need for face-mask ventilation according to the neonatal algorithm
Supplemental oxygen in delivery room | 30 minutes
  Number (percentage) of infants who needed supplemental oxygen in delivery room
Admission to the special care unit | 30 minutes
  Number (percentage) of infants who were admitted to the special care unit
Local lesions | 10 minutes
  Number (percentage) of local lesions (defined as bleeding from the mouth and/or the nose) due to suctioning procedure
Respiratory distress during the first 48 hours of life | 48 hours
  Number (percentage) of infants with respiratory distress (defined as need for supplemental oxygen and/or nasal-CPAP) during the first 48 hours of life

CONTACTS AND LOCATIONS:
Locations (1):
- St. Luke Catholic Hospital, Wolisso, Ethiopia, Addis Ababa, Ethiopia

IPD SHARING:
Plan to Share IPD: Yes
Data will be available upon reasonable request
Supporting Information: Study Protocol, SAP, ICF

REFERENCES:
- [Result] Patterson J, North K, Dempsey E, Ishoso D, Trevisanuto D, Lee AC, Kamath-Rayne BD; Newborn Brain Society Guidelines and Publications Committee. Optimizing initial neonatal resuscitation to reduce neonatal encephalopathy around the world. Semin Fetal Neonatal Med. 2021 Aug;26(4):101262. doi: 10.1016/j.siny.2021.101262. Epub 2021 Jun 22. PMID 34193380
- [Result] Foster JP, Dawson JA, Davis PG, Dahlen HG. Routine oro/nasopharyngeal suction versus no suction at birth. Cochrane Database Syst Rev. 2017 Apr 18;4(4):CD010332. doi: 10.1002/14651858.CD010332.pub2. PMID 28419406
- [Result] Lawn JE, Blencowe H, Oza S, You D, Lee AC, Waiswa P, Lalli M, Bhutta Z, Barros AJ, Christian P, Mathers C, Cousens SN; Lancet Every Newborn Study Group. Every Newborn: progress, priorities, and potential beyond survival. Lancet. 2014 Jul 12;384(9938):189-205. doi: 10.1016/S0140-6736(14)60496-7. Epub 2014 May 19. PMID 24853593
- [Result] Kamath-Rayne BD, Berkelhamer SK, Kc A, Ersdal HL, Niermeyer S. Neonatal resuscitation in global health settings: an examination of the past to prepare for the future. Pediatr Res. 2017 Aug;82(2):194-200. doi: 10.1038/pr.2017.48. Epub 2017 May 24. PMID 28419084
- See also: Related Info — http://www.helpingbabiesbreathe.org